CLINICAL TRIAL: NCT01074593
Title: Clinical Study of Pharmacokinetics and Pharmacodynamics of the Drug Interferon Beta-1a Produced By Laboratorio Quimico Farmaceutico Bergamo Compared To Interferon Beta-1a (Rebif - Merck Serono) In Healthy Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics of the Interferon Beta-1a Produced by Laboratorio Quimico Farmaceutico Bergamo Compared to Interferon Beta-1a (Rebif - Merck Serono) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: INTBER0609; VERSION 3
Record Dates: First submitted 2009-11-13; First posted 2010-02-24 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: PHARMACOKINETICS AND PHARMACODYNAMICS OF DRUG INTERFERON BETA-1A
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Bergamo - Interferon beta-1a
  Interventions: Biological: Interferon beta-1a
- Comparator - Merck Serono (Active Comparator): Merck Serono - Interferon beta-1a
  Interventions: Biological: Interferon beta-1a

INTERVENTIONS:
Biological: Interferon beta-1a — 12.000UI - single dose
  Arms: Test
Biological: Interferon beta-1a — 12.000UI - Single dose
  Arms: Comparator - Merck Serono

SUMMARY:
The primary objective of this study is to compare the pharmacokinetic and pharmacodynamic effect of two commercial preparations of interferon beta-1a (IFN Test: Lab Bergamo and IFN Comparator: Rebif ® - Merck Serono Lab) after single administration (12.000UI) in healthy subjects by modifying the parameters Cmax, Tmax and AUC (pharmacokinetics) and the levels of 2'5' oligoadenylate synthase and beta-2-microglobulin (pharmacodynamics).

DETAILED DESCRIPTION:
Secondly, safety will be observed (tolerability) clinically after administration of a single dose in study subjects, by comparing the clinical and laboratory parameters before and after study and the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Accepted Informed Consent
2. Study subjects male, aged 18 to 50 years;
3. Research subjects with body mass index greater than or equal to 19 and less than or equal to 30;
4. Subjects considered healthy, based on the analysis of the clinical history and clinical and laboratory data.

Exclusion Criteria:

1. Having donated or lost 450 mL or more of blood in the 6 months preceding the study;
2. Have participated in any experimental study or have ingested any drug trial in the 12 months preceding the start of the study;
3. Having made regular use of medication in the 4 weeks prior to the start of the study or have made use of medications that interfere with the pharmacokinetics / pharmacodynamics of drugs studied a week before the start of the study;
4. Have been hospitalized for any reason, up to 8 weeks before the start of the study;
5. Demonstrate a history of alcohol abuse, drugs, or drugs, or have consumed alcohol within 48 hours prior to the period of hospitalization;
6. Have a history of liver disease, renal, pulmonary, gastrointestinal, hematological or psychiatric;
7. To present the pressure of any etiology requiring pharmacological treatment;
8. Display history of myocardial infarction, angina and / or heart failure.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Comparison of pharmacokinetic and pharmacodynamic effect between two commercial preparations of interferon beta-1a. | 168 hours
  Assessment of pharmacodynamics: cholinesterase activity 2'5' oligoadenylate synthase and beta-2-microglobulin.Pharmacokinetics measured through plasma quantification

SECONDARY OUTCOMES:
Security: observation of adverse effects | 168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil